CLINICAL TRIAL: NCT06098430
Title: A Pilot Study of Prospective Patient-Reported Outcomes and Quality of Life in Adult and Pediatric Patients With Nodular Lymphocyte-Predominant Hodgkin Lymphoma (NLPHL)
Brief Title: Patient-Reported Outcomes and Quality of Life in Adult and Pediatric Patients With Nodular Lymphocyte-Predominant Hodgkin Lymphoma (NLPHL)
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NLPHLPRO; NCI-2023-08916 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Nodular Lymphocyte-Predominant Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is a pressing need to measure patient-reported symptoms in patients of all ages diagnosed with nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL). This study aims to measure longitudinal symptom burden and treatment tolerability utilizing validated patient-reported outcomes (PROs) instruments.

Primary Objective:

* To develop the data collection infrastructure required to prospectively collect longitudinal electronic patient-reported outcomes (PROs) survey instruments in adult and pediatric patients diagnosed with NLPHL.

Secondary Objective:

* To examine differences in baseline and longitudinal changes in PROs based on disease characteristics, disease status, and treatment strategies among adult and pediatric patients diagnosed with NLPHL.

DETAILED DESCRIPTION:
The broad aim of this study is to develop the foundational data management infrastructure required to prospectively collect longitudinal electronic patient-reported outcomes (PROs) survey instruments in adult and pediatric patients diagnosed with nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL). The study team further aims to elucidate how PROs change over time and how they may be affected by different patient, disease, and treatment characteristics.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 8 years
* Patient or their adult proxy must have verbal and written English language proficiency.
* Pathologically confirmed diagnosis of nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL); patients with evidence of transformed lymphoma at diagnosis or subsequent development of transformed lymphoma after diagnosis are eligible.
* Patients or their adult proxy must be able to provide consent.
* Patients and/or adult proxy must be able to complete electronic quality of life surveys

Exclusion Criteria

* Age 7 years or less.
* Patient or adult proxy does not have verbal and written English language proficiency.
* Patients with histologic evidence of a composite lymphoma (NLPHL with a concurrent diagnosis of Hodgkin lymphoma, indolent non-Hodgkin lymphoma, or gray zone lymphoma) at diagnosis are not eligible.
* Inability or unwillingness of research participant or legal guardian/representative to give consent.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that meet eligibility
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Estimates of response rates | At baseline, 3, 6, 9, and 12 months
  Percentage of survey completion at different timepoints
Patterns of individual per-patient survey completion | At baseline, 3, 6, 9, and 12 months
  Patterns of individual per-patient survey completion will be described. Non-responders, late responders, and patients with suboptimal item completion rates who require real-time outreach will be queried for individual challenges in completing PRO surveys for iterative improvements to infrastructure.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Crabtree, PhD, Principal Investigator — St. Jude Children's Research Hospital; Ajay Major, MD, MBA, Principal Investigator — University of Colorado, Denver; Anna Jones, PhD, Principal Investigator — St. Jude Children's Research Hospital; Matthew Rees, MD, Principal Investigator — St. Jude Children's Research Hospital; Jamie Flerlage, MD, MS, Principal Investigator — University of Rochester
Locations (5):
- United States (5):
  - University of Colorado Hospital, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Rochester Medical Center, Rochester, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols